CLINICAL TRIAL: NCT01917669
Title: A Pilot Feasibility Study of Fibroblast Calcium and Glucoregulation in Health
Brief Title: A Pilot Feasibility Study of Fibroblast Calcium and Glucoregulation in Health and Disease
Status: Withdrawn | Type: Observational
Why Stopped: Funding was never available to conduct the proposed series of experiments.
Sponsor: University of Kentucky (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Olivier Thibault, PhD, Principal Investigator, University of Kentucky
Other Study IDs: 13-0571-F1V
Record Dates: First submitted 2013-07-31; First posted 2013-08-07 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and tissue (skin biopsy)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lean Non-Diabetic Group: Variables measured will also include serum analyses (HbA1c, adiponectin, cholesterol) and patient vital signs.
- Pre-diabetics: These patients are anticipated to have elevated BMI, yet not be diabetics.
- Diabetic Patients: These patients will have good glucose control.
- Diabetic patients with poor glucocontrol: These patients are anticipated to have poor glucose control. They are usually taking insulin.

SUMMARY:
The purpose of this research is to better understand how calcium and glucose may play a role in people developing diabetes. By doing this study, the investigator hopes to learn whether abnormal calcium and glucose responses in skin biopsies from healthy patients and patients with Type 2 diabetes can identify and predict patients at greatest risk for later complications.

DETAILED DESCRIPTION:
The overall goal of this proposal is to establish a pathophysiological index of a patient's status through imaging of calcium and glucose in skin fibroblasts. The investigator will obtain skin samples from patients in the Barnstable Brown Obesity and Diabetes Center at the University of Kentucky to test the hypothesis that calcium and glucose dysregulation are present in fibroblasts from patients with Type 2 diabetes, and are exaggerated in more difficult-to-treat patients or those with poor glucose control. The innovation of the project focuses on results that can potentially lead to earlier treatment for patients with diabetes and thereby reduce the risk for long-term complications.

Three levels of analyses will be conducted to assess the relationship between Ca2+ and glucose homeostasis in four patient groups (lean non-diabetics, obese non-diabetics, Type 2 Diabetics with good glucose control, and Type 2 Diabetics with poor control.

Participants will be required to attend only one study visit that will last approximately 2-3 hours. During the study subject will undergo the following: 1. Collection of two 4 ml tubes of blood for adiponectin analysis, 2. A skin biopsy, 3. Collection and review of medical history and current/past medication use 4. Collection of demographic information, 5. Height and weight measurement 6. Body mass index evaluation, 7. Vital signs assessment (blood pressure, pulse).

Follow-up for all enrolled patients will occur on a yearly basis through a phone interview.

The punch biopsy will be performed under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Type 2 Diabetes

Exclusion Criteria:

* Under 40 years of age
* Over 55 years of age
* Pregnant or breastfeedig
* Will not agree to a skin biopsy
* Talking calcium channel blockers

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit both male and female participants. The age range for this study is 40-55 years old
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Are peak (nM) calcium responses to bradykinin enhanced along the continuum of disease in skin fibroblasts from the 4 patient groups? | Three years
  All participants groups will be compared statistically to the lean patient group.

SECONDARY OUTCOMES:
Are glucose utilization rates (a.u./min) measured in skin fibroblasts from the 4 patient groups different with disease progression? | Three years
  A unitless index of health status based on serum analyses (cholesterol, adiponectin, HbA1c) for each patient will be correlated with a unitless index of glucose status based on fibroblast imaging data.

OTHER OUTCOMES:
What component of peripheral metabolic dysregulation (HbA1c (%), adiponectin (ug/mL), cholesterol (mg/dL)) is associated with changes in calcium responses (nM) in skin fibroblasts? | Three years
  The investigator will also focus on two groups of patients, obese-non-diabetics and diabetics with poor control, during the analysis period and prospectively follow these patients for clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Thibault, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky Center for Clinical and Translational Science, Lexington, Kentucky, United States